CLINICAL TRIAL: NCT04595240
Title: Semen Analysis Changes in Covid-19 Positive Patients
Brief Title: Semen Analysis Changes in Covid-19 Positivepatients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mostafa kamel abdel rahman abdel aal, investigator, Assiut University
Other Study IDs: Semen analysis post covid-19
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: semen analysis — semen analysis

SUMMARY:
The viral pandemic of the coronavirus disease 2019 (COVID-19), generated by a novel mutated severe acute respiratory syndrome coronavirus (SARS-CoV-2), has become a serious worldwide public health emergency, evolving exponentially. While the main organ targeted in this disease is the lungs, other vital organs, such as the heart and kidney, may be implicated. The main host receptor of the SARS-CoV-2 is angiotensin converting enzyme 2 (ACE2), a major component of the renin-angiotensin-aldosterone system (RAAS). The ACE2 is also involved in testicular male regulation of steroidogenesis and spermatogenesis. As the SARS-CoV-2 may have the potential to infect the testis via ACE2 and adversely affect male reproductive system.

DETAILED DESCRIPTION:
A recent report published in JAMA Network Open revealed that in an analysis 38 semen samples from COVID-19 patients, 6 (four at the acute stage of infection and, alarmingly, two who were recovering) tested positive for the virus by RT-PCR.

Importantly, at this point, the investigators have no idea whether the actual virus was viable and infectious. Nevertheless, the possibility that this coronavirus could have a pathophysiological impact on the testes was suggested by additional data indicating that active COVID-19 infection dramatically reduced the testosterone-to-LH ratio, suggesting a significant impact on the responsiveness of Leydig cells to LH stimulation In many ways, the investigators should not be surprised by these observations because the blood-testes barrier is known to offer little defense against viral invasion, given the wide range of pathogenic viruses (HIV, hepatitis, mumps, papilloma) that are known to be capable of damaging the testes and rendering the host infertile.

The angiotensin system plays a critical role in the survival and functionality of human spermatozoa but also creates a vulnerability to COVID-19 attack. Angiotensin 1 is a biologically inactive decapeptide that is cleaved by ACE1 to create angiotensin II, which in turn activates the AT1R and AG2R receptors, both of which are present in these cells. Angiotensin II is further processed by ACE2 to generate angiotensin 1-7 which binds the MAS receptor activating PI3K. The latter then phosphorylates AKT, which maintains cell viability by phosphorylating key regulators of sperm apoptosis such as BAD. As long as BAD is phosphorylated, it is held in abeyance by a 14-3-3 keeper protein. However, if the PI3/AKT pathway becomes compromised, BAD dephosphorylates, is released from its association with 14-3-3, and moves to the mitochondria where it inactivates anti-apoptotic factors and promotes the intrinsic apoptotic cascade. The spike protein on COVID-19 specifically targets ACE2 and in so doing removes an important stimulus for PI3K/AKT, thereby compromising sperm viability. Subsequent to COVID-19 binding, the ectodomain of ACE2 may be removed by ADAM proteases and shed from the sperm surface. Alternatively proteases from the TMPRSS-family, either as intrinsic components of the sperm plasma membrane or delivered by seminal prostasomes, can facilitate fusion between the virus and the sperm surface by cleaving ACE2 and the viral spike proteins (S1 and S2) at the sites indicated by dashed lines, thereby completing the transformation of this cell from procreating gamete to viral vector.

An additional concern of the COVID-19 pandemic that might impact male fertility is fever. Particularly high and sustained elevation in body temperature is a major manifestation of the COVID-19 pandemic, which complicates more than 80% of patients. The concept that fever and elevation of testicular temperature result in impairment of spermatogenesis is widely accepted.

More importantly, emerging evidence indicates that a subgroup of patients with severe COVID-19 might have a secondary cytokine storm syndrome (hemophagocytic lymphohistiocytosis). This is an underrecognized, hyperinflammatory syndrome characterized by sustained fever, with fulminant and fatal hypercytokinemia with multiorgan failure. These patients have a particular serum blood cytokine profile with cytopenia and hyperferritinemia. These findings also suggest that immunomodulatory therapy (IL-6 antagonist) may improve mortality rate considerably in these patients.

As cytokines contribute to testicular function and maintenance of male reproductive health, and to the pathologies associated with their abnormal activity in this organ, COVID-19-induced changes in cytokines profile may have further implications to male fertility. In addition, immunomodulatory therapies may provoke potential long-term effects on male fertility and are a matter of concern. Furthermore, cytokine microenvironment deviations within the testis may have tumorigenic adverse effects on the cellular level, leading eventually to testicular cancer, a second long-term matter of concern.

Aim of the study :

Know the Effect of covid-19 on spermatogenesis

ELIGIBILITY:
Inclusion Criteria:

* adult male patient age younger than 45 years old
* no history of fertility disorders
* good body built and secondary sexual charcter .

Exclusion Criteria:

* congenital anomalies of the testis
* chronically ill patients
* proplems of male fertility
* males with varicocele
* sexual performance disorders .

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: men with th mentioned criteria
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
changes of semen volume in (ML)by covid-19 from normal values. | 72days after infection
  semen analysis taken by 72day of infection to see the effect on the new cycle of spermatogenesis
changes of sperm concentration in (million/ml) by covid-19 from normal values. | 72days after infection
  semen analysis taken by 72day of infection to see the effect on the new cycle of spermatogenesis
changes of sperm morphology in (percentage of normal forms) by covid-19 from normal values. | 72days after infection
  semen analysis taken by 72day of infection to see the effect on the new cycle of spermatogenesis
changes of sperm motility in percentage of (A+B) by covid-19 from normal values. | 72days after infection
  semen analysis taken by 72day of infection to see the effect on the new cycle of spermatogenesis
changes of semen volume in (ML) by covid-19 from from the first sample | after 72 days of the first sample
  semen analysis taken by 72day of the first negative swab of covid-19 to see the effect on the new cycle of spermatogenesisand to compare with the first sample which done during infection.
changes of sperm concentration in (million /ML) by covid-19 from from the first sample | after 72 days of the first sample
  semen analysis taken by 72day of the first negative swab of covid-19 to see the effect on the new cycle of spermatogenesisand to compare with the first sample which done during infection.
changes of sperm morphology in percentage of normal form by covid-19 from from the first sample | after 72 days of the first sample
  semen analysis taken by 72day of the first negative swab of covid-19 to see the effect on the new cycle of spermatogenesisand to compare with the first sample which done during infection.
changes of sperm motility in percentage of (A+B) by covid-19 from from the first sample | after 72 days of the first sample
  semen analysis taken by 72day of the first negative swab of covid-19 to see the effect on the new cycle of spermatogenesisand to compare with the first sample which done during infection.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed a abdel moniem, md, Study Director — Assiut University
Locations (1):
- Mostafa Kamel, Asyut, Egypt

REFERENCES:
- [Derived] Mohammed N, Kamel M, Gadelkareem RA, Zarzour MA, Kurkar A, Abdel-Moniem AM, Behnsawy H. Semen quality changes during infection and recovery phases of mild-to-moderate COVID-19 in reproductive-aged patients: a prospective case series. Basic Clin Androl. 2023 Jan 19;33(1):2. doi: 10.1186/s12610-022-00175-7. PMID 36653786